CLINICAL TRIAL: NCT04789525
Title: Clinical (BMI & MRI) and Biochemical (Adiponectin, Leptin, TNF-α & IL-6) Effects of High-intensity Aerobic Training With High Protein Diet in Childhood Obesity Following COVID-19 Infection
Brief Title: Physical Training and Diet for Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Obesity
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (high-intensity aerobic training with high protein diet ) (Experimental)
  Interventions: Other: High-intensity aerobic training with high protein diet
- Group B(regular physical activities and taken regular diet) (Experimental)
  Interventions: Other: High-intensity aerobic training with high protein diet

INTERVENTIONS:
Other: High-intensity aerobic training with high protein diet — High-intensity aerobic training was given with 50 to 70 % of the maximum heart rate. the intervention started with 10 mins of warm-up exercise through stretching of upper and lower limb muscles. Subsequent to stretching, the subjects were asked to do 30 mins of exercises; consisting of 20 mins on the treadmill and 10 mins of cycle ergometer at 50 to 70 % of MHR, then with 10 mins of cool down.

SUMMARY:
It is observed that children affected with COVID-19 who are physically inactive or in a sedentary lifestyle may induce and develop childhood obesity (CO). the management of this clinical condition has received very little attention, there is no well-defined exercise protocols or dietary prescription for this special population; therefore, it needs an elaborative trial in this field, so the aim of his study was to find the clinical and biochemical effects of high-intensity aerobic training with a high protein diet in childhood obesity following COVID-19 infection

ELIGIBILITY:
Inclusion Criteria:

* A positive diagnosis of COVID-19
* Male children
* 5 - 12 years of age Body mass index (BMI).
* Between 85t h to 99th percentiles were considered for childhood obesity.

Exclusion Criteria:

* Subjects with a history of physical training
* Taking medications, recent surgeries.
* Fractures and joint problems in the lower extremity.
* Cardiac and respiratory problems.
* Neurological issues, major psychiatric problems.
* Any other systemic diseases, contraindications for physical training.

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male children.
Enrollment: 76 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Body mass index | 6 monthes
  For children, age adjusted BMI percentile (BMI %) was calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No